CLINICAL TRIAL: NCT07044193
Title: Reversal of Pipecuronium-induced Neuromuscular Blockade With Sugammadex During Sevoflurane Anesthesia: a Drug Safety Randomised Controlled Trial
Brief Title: Reversal of Pipecuronium-induced Neuromuscular Blockade With Sugammadex During Sevoflurane Anesthesia
Acronym: RPINMBWS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, MD PhD, University of Debrecen
Organization: University of Debrecen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AITT 2025/2; DE RKEB/IKEB 7108-2025 (Other: Regional and Institutional Ethics Committee University of Debrecen Clinical Center); NNGYK/ETGY/08365-4/2025 (Other: National Center for Public Health and Pharmacy Department of Clinical Research)
Record Dates: First submitted 2025-06-19; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Neuromuscular Blocking Agents; Residual Neuromuscular Block; Reversal of Neuromuscular Blockade
Keywords: reversal of neuromuscular blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Pipecuronium; Rocuronium

STUDY DESIGN:
Intervention Model Description: controlled, randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rocuronium bromide as a control muscle relaxant agent in comparison to pipecuronium bromide. (Active Comparator): Rocuronium bromide induced neuromuscular blockade antagonised by sugammadex as a control.
  Interventions: Drug: Rocuronium bromide
- Reversal of pipecuronium induced neuromuscular blockade using sugammadex. (Experimental): Reversal of pipecuronium induced neuromuscular blockade using sugammadex.
  Interventions: Drug: pipecuronium bromide

INTERVENTIONS:
Drug: pipecuronium bromide — Investigation of muscle relaxation with pipecuronium bromide
  Arms: Reversal of pipecuronium induced neuromuscular blockade using sugammadex.
Drug: Rocuronium bromide — Muscle relaxation with rocuronium as a control
  Arms: Rocuronium bromide as a control muscle relaxant agent in comparison to pipecuronium bromide.

SUMMARY:
Safety during modern practice of anaesthesia is of great concern. Patients admitted daily for surgical procedures undergoing general anaesthesia for different types of operations are exposed to different risks, starting from the anaesthesia and ending with the surgical intervention. Aim of the study is to provide a comprehensive and evidence based data regarding the safety of the neuromuscular blocking agents used in modern anaesthesia practice, precisely Rocuronium and Pipecuronium, as well as the reversal agents such as Sugammadex, which is the sole agent in use in practice nowadays. A routine anaesthetic practice will be performed during the whole period of our study after strict patient selection criteria. Intraoperative standard monitoring as per local and international guidelines will be applied, this includes Spo2, ECG, NIBP/IBP, etCO2, BIS and Tetragaph for neuromuscular blockade monitoring. After induction of anaesthesia and prior to the administration of the muscle relaxant agent, a TOFC (Train of Four Count) will be registered as the starting point. Throughout the anaesthetic time, there will be continuous TOF monitoring. The anaesthesia will be maintained by sevoflurane. Also, the recruited samples will be divided according to the neuromuscular blockade agents administered, either Rocuronium or Pipecuronium. At the end of the surgical procedure, the time lapse between the administration of the reversal agent Sugammadex and a TOF ratio of 0.9 is registered as our primary end point. TOF measures will be performed in the postoperative period, to make sure there is no residual neuromuscular blockade in the early postoperative phase. The study will not only monitor the safety of the neuromuscular blocking agents in use, but will also monitor any signs of anaphylaxis due to their administration both intra and postoperatively.

DETAILED DESCRIPTION:
Pipecuronium bromide (Arduan®) is a long-acting (45-100 min) aminosteroid-type muscle relaxant which has no cardiovascular side effects, neither causes histamine release and it is primarily excreted from the body via the liver and partially via the kidney. These properties make it the drug of choice Pipecuronium in long (≥100 min) operations and intensive care units. Currently, it is the only available long acting muscle relaxant in Hungary. Pipecuronium is also licensed and used regularly in other countries as per (www.drugs.com/international). Residual neuromuscular blockade is considered a characteristic of the long-acting muscle relaxants, which in turn could lead to postoperative respiratory complications.

Therefore, adequate reversal of pipucornium induced neuromuscular blockade is crucial as a patient safety criterion.

Neuromuscular block reversal using neostigmine has proved to be non-reliable. There is a good evidence of the risks and inadequacy of neostigmine reversal, particularly in the case of inhalational anaesthetics . Therefore, the use of a more effective and safe antagonist may offer significant advantages in the use of Pipecuronium and open a new perspective in neuromuscular blockade reversal. Sugammadex (Bridion®) is the first muscle relaxant antagonist to bind and neutralise muscle relaxants in the plasma. The cyclodextrin compound was originally developed to antagonize Rocuronium block, but it is also able to reverse the Vecuronium bromide-induced block, due to structure similarity. Sugammadex binds to Pipecuronium bromide, which also has an aminosteroid structure, and has an affinity for it that is about ten times that of Rocuronium bromide http://www.pmda.go.jp/files/000153538.pdf. Several studies have demonstrated the efficacy of Sugammadex in antagonizing Rocuronium-induced neuromuscular block, but in the international literature, few clinical data are available regarding the safety of Sugammadex as a reversal agent for Pipecuronium blockade. In a previous study was found that Sugammadex also antagonizes the residual effect of Pipecuronium when neuromuscular blockade already shows signs of spontaneous recovery: two muscle twitches (moderate, so-called TOF-Count 2 block) can be elicited by Train-of-Four (TOF) stimulation. Sugammadex at a relatively low dosage (1 mg/kg) was sufficient to achieve adequate effects in patients with moderate Pipecuronium-induced blockade (TOFC2). There was no postoperative muscle weakness or recurrence encountered. It was demonstrated that 2 mg/kg sugammadex can effectively reverse Pipecuronium-induced deep neuromuscular block. In this study, was also demonstrated that neither residual nor recurreIt that muscle relaxant effects should arise after antagonizing deep Pipecuronium block with Sugammadex .

Allergic reactions may occur with the use of muscle relaxants. While Rocuronium bromide is the second most common cause anaphylactic reactions among muscle relaxants in use, which is not revealed in the case of Pipecuronium. No large case-control studies have yet been performed to investigate the safety of reversing Pipercuornium-induced blockade using Sugammadex, neither the incidence of postoperative residual neuromuscular block, nor the incidence of anaphylactic reactions post-administration.

The aim of present study is therefore to investigate the safety of Pipecuronium in comparison to Rocuronium bromide in surgical patients' population undergoing anaesthesia with sevoflurane. The study will evaluate the effective reversing ability of Sugammadex, assessing the incidence of postoperative residual neuromuscular block and the incidence of allergic reactions, nevertheless comparing different doses of sugammadex required to antagonise the effects of the two muscle relaxants.

ELIGIBILITY:
Inclusion Criteria:

* 80 adult general surgery and neurosurgical patients are enrolled in the study after giving an informed written consent regarding their participation.
* Age: between 18-65 years;
* ASA score: 1-3;
* BMI 18.5-25 (normal body weight);
* Males and females were recruited in an equal ratio;
* Minimal surgical time of at least ≥ 40 minutes;
* Procedures requiring endotracheal intubation;

Exclusion Criteria:

* Diseases affecting neuromuscular function (myopathies, severe liver and kidney failure);

  * Drugs affecting neuromuscular function (magnesium, aminoglycosides);
  * Difficult airway, or anticipated difficult intubation;
  * Pregnancy (a pregnancy test is performed in women of childbearing age to rule out pregnancy);
  * Breast-feeding;
  * Acute surgery;
  * COPD
  * Glaucoma
  * History of previous allergic/anaphylactic reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-26 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time till TOF ratio of 0.9 | from reversal to extubation within 5 minutes as per the onset of time of Sugammadex
  The time between the start of sugammadex administration and reaching a TOF ratio of 0.9 will be the primary efficacy endpoint of the study.

SECONDARY OUTCOMES:
Incidence of residual neuromuscular blockade | 30 minutes after extubation
  The Prevalence of TOF <0.9 in the postoperative period.

OTHER OUTCOMES:
The incidence of allergic/anaphylactic reactions | From induction to up to 30 minutes postoperatively
  The incidence of allergic/anaphylactic reactions associated with muscle relaxant and reversal agents' administration.
Time to achieving a TOF ratio of 1.0 | the time elapsed until the onset of Summadex which is within 5 minutes
  The time elapsed between Sugammadex administration and achieving a TOF ratio of 1.0
Doses of the muscle ralaxants | from induction to reversal according to the surgical time
  Comparison of sugammadex doses required to reverse the effects of the study focused two muscle relaxants.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naguib M, Brull SJ, Kopman AF, Hunter JM, Fulesdi B, Arkes HR, Elstein A, Todd MM, Johnson KB. Consensus Statement on Perioperative Use of Neuromuscular Monitoring. Anesth Analg. 2018 Jul;127(1):71-80. doi: 10.1213/ANE.0000000000002670. PMID 29200077
- [Background] Cardona V, Ansotegui IJ, Ebisawa M, El-Gamal Y, Fernandez Rivas M, Fineman S, Geller M, Gonzalez-Estrada A, Greenberger PA, Sanchez Borges M, Senna G, Sheikh A, Tanno LK, Thong BY, Turner PJ, Worm M. World allergy organization anaphylaxis guidance 2020. World Allergy Organ J. 2020 Oct 30;13(10):100472. doi: 10.1016/j.waojou.2020.100472. eCollection 2020 Oct. PMID 33204386
- [Background] Fuchs-Buder T, Brull SJ, Fagerlund MJ, Renew JR, Cammu G, Murphy GS, Warle M, Vested M, Fulesdi B, Nemes R, Columb MO, Damian D, Davis PJ, Iwasaki H, Eriksson LI. Good clinical research practice (GCRP) in pharmacodynamic studies of neuromuscular blocking agents III: The 2023 Geneva revision. Acta Anaesthesiol Scand. 2023 Sep;67(8):994-1017. doi: 10.1111/aas.14279. Epub 2023 Jun 22. PMID 37345870
- [Background] Samuel WM, Holmes JC. Search for elaphostrongyline parasites in cervids from Alberta. Can J Zool. 1974 Mar;52(3):401-3. doi: 10.1139/z74-048. No abstract available. PMID 4819478
- [Background] Tassonyi E, Asztalos L, Szabo-Maak Z, Nemes R, Pongracz A, Lengyel S, Fulesdi B. Reversal of Deep Pipecuronium-Induced Neuromuscular Block With Moderate Versus Standard Dose of Sugammadex: A Randomized, Double-Blind, Noninferiority Trial. Anesth Analg. 2018 Dec;127(6):1344-1350. doi: 10.1213/ANE.0000000000003719. PMID 30169407
- [Background] Tassonyi E, Pongracz A, Nemes R, Asztalos L, Lengyel S, Fulesdi B. Reversal of Pipecuronium-Induced Moderate Neuromuscular Block with Sugammadex in the Presence of a Sevoflurane Anesthetic: A Randomized Trial. Anesth Analg. 2015 Aug;121(2):373-80. doi: 10.1213/ANE.0000000000000766. PMID 25923435
- [Background] Pongracz A, Szatmari S, Nemes R, Fulesdi B, Tassonyi E. Reversal of neuromuscular blockade with sugammadex at the reappearance of four twitches to train-of-four stimulation. Anesthesiology. 2013 Jul;119(1):36-42. doi: 10.1097/ALN.0b013e318297ce95. PMID 23665915
- [Background] Puhringer FK, Gordon M, Demeyer I, Sparr HJ, Ingimarsson J, Klarin B, van Duijnhoven W, Heeringa M. Sugammadex rapidly reverses moderate rocuronium- or vecuronium-induced neuromuscular block during sevoflurane anaesthesia: a dose-response relationship. Br J Anaesth. 2010 Nov;105(5):610-9. doi: 10.1093/bja/aeq226. Epub 2010 Sep 28. PMID 20876699
- [Background] Duvaldestin P, Kuizenga K, Saldien V, Claudius C, Servin F, Klein J, Debaene B, Heeringa M. A randomized, dose-response study of sugammadex given for the reversal of deep rocuronium- or vecuronium-induced neuromuscular blockade under sevoflurane anesthesia. Anesth Analg. 2010 Jan 1;110(1):74-82. doi: 10.1213/ANE.0b013e3181c3be3c. Epub 2009 Nov 21. PMID 19933538
- [Background] Suy K, Morias K, Cammu G, Hans P, van Duijnhoven WG, Heeringa M, Demeyer I. Effective reversal of moderate rocuronium- or vecuronium-induced neuromuscular block with sugammadex, a selective relaxant binding agent. Anesthesiology. 2007 Feb;106(2):283-8. doi: 10.1097/00000542-200702000-00016. PMID 17264722
- [Background] Abrishami A, Ho J, Wong J, Yin L, Chung F. Cochrane corner: sugammadex, a selective reversal medication for preventing postoperative residual neuromuscular blockade. Anesth Analg. 2010 Apr 1;110(4):1239. doi: 10.1213/ANE.0b013e3181ce8d5e. PMID 20357160
- [Background] Kirkegaard H, Heier T, Caldwell JE. Efficacy of tactile-guided reversal from cisatracurium-induced neuromuscular block. Anesthesiology. 2002 Jan;96(1):45-50. doi: 10.1097/00000542-200201000-00013. PMID 11753000
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20357160/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11753000/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17264722/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19933538/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20876699/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23665915/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25923435/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30169407/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/4819478/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37345870/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33204386/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29200077/
- Available data/document: Study Protocol — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2025-521375-31-00